CLINICAL TRIAL: NCT01497769
Title: A Phase I Trial to Compare the Safety and Immunogenicity of Candidate TB Vaccine MVA85A Administered by the Aerosol Inhaled Route and the Intradermal Route in Healthy BCG-vaccinated Adult Subjects
Brief Title: Safety of Tuberculosis Vaccine, MVA85A, Administered by the Aerosol Route and the Intradermal Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TB026
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Tuberculosis
Keywords: vaccine; immunogenicity
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Aerosol inhaled MVA85A and intradermal saline placebo
  Interventions: Biological: Aerosol inhaled MVA85A
- Group 2 (Experimental): Intradermal MVA85A and inhaled aerosol saline placebo
  Interventions: Biological: Intradermal MVA85A

INTERVENTIONS:
Biological: Aerosol inhaled MVA85A — Aerosol inhaled MVA85A 1 x 10^7 pfu and intradermal saline placebo
  Arms: Group 1
Biological: Intradermal MVA85A — Intradermal MVA85A 1 x 10^7 pfu and inhaled aerosol saline placebo
  Arms: Group 2

SUMMARY:
This is a phase I trial to compare the safety and immunogenicity of candidate TB vaccine MVA85A administered by the aerosol inhaled route and the intradermal route in healthy BCG-vaccinated adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-50 years
* Resident in or near Oxford for the duration of the trial period
* No relevant findings in medical history or on physical examination
* Confirmation of prior vaccination with BCG not less than 6 months prior to projected trial vaccination date (by visible BCG scar on examination or written documentation)
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register subject details with a confidential database to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

* Any respiratory disease, including asthma
* Current smoker
* Clinically significant abnormality on screening chest x rays
* Clinically significant abnormality of pulmonary function tests
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Current use of any medication taken through the nasal or inhaled route including cocaine or other recreational drugs
* Laboratory evidence at screening of latent M.tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Previous vaccination with candidate vaccine MVA85A or candidate vaccine FP85A or any other recombinant MVA vaccine
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine, sedative drugs, or any local or general anaesthetic agents
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the subject in the trial
* Positive HBsAg, HCV or HIV antibodies
* Female currently lactating, confirmed pregnancy or intention to become pregnant during trial period
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the trial vaccine for 30 days prior to dosing with the trial vaccine, or planned use during the trial period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the subject at risk or may influence the result of the trial or may affect the subject's ability to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety of MVA85A vaccination by the aerosol inhaled route | 24 weeks following vaccination
  To evaluate the safety in healthy BCG-vaccinated subjects of MVA85A vaccination by the aerosol inhaled route by actively and passively collecting data on adverse events

SECONDARY OUTCOMES:
Immunogenicity of MVA85A vaccination by the aerosol inhaled route compared with the intradermal route | 24 weeks following vaccination
  To evaluate the systemic and mucosal cellular immunogenicity in healthy BCG-vaccinated subjects of MVA85A vaccination by the aerosol inhaled route compared with the intradermal route by comparing laboratory markers of cell mediated immunity in blood and bronchoalveolar lavage samples

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- Centre of Clinical Vaccinology and Tropical Medicine (CCVTM) Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Satti I, Meyer J, Harris SA, Manjaly Thomas ZR, Griffiths K, Antrobus RD, Rowland R, Ramon RL, Smith M, Sheehan S, Bettinson H, McShane H. Safety and immunogenicity of a candidate tuberculosis vaccine MVA85A delivered by aerosol in BCG-vaccinated healthy adults: a phase 1, double-blind, randomised controlled trial. Lancet Infect Dis. 2014 Oct;14(10):939-46. doi: 10.1016/S1473-3099(14)70845-X. Epub 2014 Aug 20. PMID 25151225